CLINICAL TRIAL: NCT05527847
Title: A Pilot Randomized Clinical Trial (RCT) to Examine the Benefits of a Culturally Adapted Peer Support and Self-Management Intervention to Improve Glycemic Control in African Americans
Brief Title: Peers EXCEL Trial to Improve Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-0879; A561000 (Other: UW Madison); PHARM/PHARMACY (Other: UW Madison); Protocol Version 02/20/2023 (Other: UW Madison)
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes
Keywords: African-American; medication adherence; diabetes self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Living with Diabetes (HLWD) (Active Comparator): Participants will have a 6-week self-management program, followed by the option to work with a Community Health Worker for the remaining 4 months.
  Interventions: Behavioral: HLWD
- Peers EXCEL (Experimental): Participants will have an 8-week self-management program, and will participate in phone calls with a peer for the remaining 4 months.
  Interventions: Behavioral: Peers LEAD; Behavioral: HLWD

INTERVENTIONS:
Behavioral: Peers LEAD — Two group session focusing on beliefs about medicines and diabetes, discrimination/mistrust, and communication with providers, and 2 peer-based phone calls from Ambassadors to occur weekly for weeks 3-8, then bi-weekly for weeks 9-12.
  Arms: Peers EXCEL
Behavioral: HLWD — Weekly group sessions for two months. Sessions will last up to 2.5 hours and focus on a different diabetes self-management topic.

SUMMARY:
The purpose of the study is to gather input about the value of adding a newly developed diabetes self-management program to an existing diabetes self-management program. Participants will self-identify as African-American/Black with type 2 diabetes, and prescribed a diabetes medication. Participants can expect to be in the study for 6 months.

DETAILED DESCRIPTION:
Both programs utilized in this study focus on topics such as diet, exercise, and stress. Both programs offer ideas to manage diabetes symptoms, discuss appropriate exercises, provide guidance on healthy eating, review the use of medicine, and offer tips on communicating with healthcare providers and voicing concerns to family members.

The new program is culturally-tailored for African Americans and focuses on helping patients take their medicines as prescribed.

The purpose of this research study is to evaluate this newly developed combined diabetes self-management program.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-90 years old
* Self-identify as African-American
* Diagnosis of Type 2 diabetes
* Able to speak/read English
* Self-report having a primary care provider who prescribes one diabetes medication
* Diagnosed with diabetes for ≥1 year at point of care
* Will reside in the geographical area throughout the study period
* Self-reported nonadherence on the DOSE-nonadherence survey
* ≥7.5% A1C

Exclusion Criteria:

* Self-reported bipolar or personality disorders, schizophrenia, Alcohol and Other Drug Abuse (AODA), dementia
* Older adults who have a history of severe hypoglycemia requiring medical assistance or glucagon administration
* Participating in another lifestyle or medication adherence program

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose (hemoglobin A1C) | Baseline, 2 months, 6 months
  The hypothesis is that there will be a more significant change in mean A1C, which is clinically meaningful, for participants in Peers EXCEL as compared to those in HLWD.

SECONDARY OUTCOMES:
Medication adherence | Baseline, 2 months, 6 months
  The hypothesis is that there will be higher medication adherence for participants in Peers EXCEL as compared to those in HLWD. Self-reported medication adherence is measured using the 3-item Extent of Nonadherence domain in the Domains of Subjective Extent of Nonadherence (DOSE-Nonadherence) survey. This measure screens for nonadherence and is calculated by computing the mean of the 3 items (range of score is 1-5). Mean scores of 3 (i.e., scoring "1" on each of the 3 items) will be classified as nonadherent, while all mean scores >3 will be classified as adherent.
Feasibility of intervention | Baseline, 2 months, 6 months
  Participants will complete validated surveys to assess diabetes-health beliefs, patient self-efficacy/activation, and patient-provider communication quality.
Acceptability of intervention | Baseline, 2 months, 6 months
  Interviews and focus groups will be conducted with participants, ambassadors and HLWD leaders respectively to get feedback on their intervention experiences.
Adherence to Refills and Medicines Scale for Diabetes (ARMS-D) Score | Baseline, 2 months, 6 months
  The ARMS-D has a total possible range of scores from 11-44, with higher scores indicating increased problems with medication adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Olayinka Shiyanbola, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No